CLINICAL TRIAL: NCT00194324
Title: Vaginal Imaging Study to Evaluate the Effect of Exercise on the Distribution of Miconozole Nitrate OVULE
Brief Title: Effect of Exercise on Spread of the Miconozole Nitrate OVULE in the Vagina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Kurt T Barnhart, MD, MSCE, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 708889; RRU010
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Health; Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Miconazole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Miconazole nitrate
Procedure: Magnetic resonance imaging
Behavioral: Moderate levels of exercise

SUMMARY:
This study uses MRI to detect the spread of the Miconozole Nitrate OVULE within the vagina. The effect of moderate amounts of physical activity on the spread will be evaluated, and compared to no physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Not at risk for pregnancy
* Willing to abstain from intercourse 24 hours prior to MRI
* Regular menstrual cycles (every 23-38 days)
* At least 10 weeks from most recent pregnancy outcome and had 2 spontaneous menstrual cycles since
* Normal pap smear within previous 12 months
* Negative test for yeast, bacterial vaginosis and trichomonas
* Not allergic to any component of the formulation
* No contraindications to MRI
* Not participated in another investigational trial within 30 days
* No history of condition, or finding on exam, that, in the opinion of the investigator, would make participation unsafe for the volunteer or complicate interpretation of the data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2004-07; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
To compare between exercise and no exercise:
Time needed for the capsule to dissolve;
Quantify and describe product distribution at 20 minute intervals within the first 90 minutes after insertion;
Quantify systemic levels of miconozole nitrate 90 minutes and 24 hours after insertion;
Quantify amount of miconozole nitrate in the vagina 90 minutes and 24 hours after insertion

SECONDARY OUTCOMES:
Product distribution will be assessed by:
Linear spread from the cervix covered by the product;
Percent of maximal linear spread from the cervix;
Surface area covered by the product;
Percent of maximal surface contact;
Presence bare spots in coating;
Presence of product outside the introitus

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States